CLINICAL TRIAL: NCT00783133
Title: Preference Evaluation of Clarinex Tablets vs. Allegra Tablets in Subjects With Symptomatic Seasonal Allergic Rhinitis
Brief Title: Preference for Clarinex Tablets vs. Allegra Tablets in Patients With Seasonal Allergies (Study P03177)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P03177
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — desloratadine; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarinex followed by Allegra (Experimental): Clarinex 5 mg by mouth daily for 7 days followed by Allegra 180 mg by mouth daily for 7 days, with 5-28 days washout between treatments.
  Interventions: Drug: Desloratadine 5 mg; Drug: fexofenadine
- Allegra followed by Clarinex (Experimental): Allegra 180 mg by mouth daily for 7 days followed by Clarinex 5 mg by mouth daily for 7 days, with 5-28 days washout between treatments.
  Interventions: Drug: Desloratadine 5 mg; Drug: fexofenadine

INTERVENTIONS:
Drug: Desloratadine 5 mg — Clarinex 5 mg daily x 7 days
  Other Names: Clarinex, SCH 034117
Drug: fexofenadine — Allegra 180 mg daily x 7 days
  Other Names: Allegra®

SUMMARY:
This was a crossover study designed to see if patients with seasonal allergy symptoms preferred Clarinex® or Allegra®. Patients were randomized to take 7 days of Clarinex or Allegra treatment, followed by a 5 to 28-day washout period (days when no drug is given), followed by 7 days of the opposite treatment. At the end of each 7-day treatment, patients were asked questions to determine which drug, Clarinex or Allegra, the patient prefers more.

ELIGIBILITY:
Inclusion Criteria:

* had at least a two-year history of seasonal allergic rhinitis;
* currently experiencing symptoms of SAR, including nasal symptoms at Visits 2 and 4, prior to entering each treatment phase;
* had not taken Allegra® or Clarinex® within the previous year;
* were 18 years of age or older;
* had negative urine test (hCG) for females of childbearing potential;
* for women of childbearing potential, agreed to use a medically accepted method of birth control;
* were free of any clinically significant disease (other than SAR) that would interfere with study evaluations;

Exclusion Criteria:

* were pregnant or nursing;
* had allergic or idiosyncratic reaction to antihistamines;
* had current or history of frequent, clinically significant sinusitis or chronic purulent nasal discharge;
* had rhinitis medicamentosa or nasal structural abnormalities (including large nasal polyps and marked septal deviation) that significantly interfered with nasal airflow;
* in the opinion of the Investigator, were dependent upon nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids (ie., subjects who could or would not observe the washout period for these prohibited medications);
* had an upper respiratory tract or sinus infection that required antibiotic therapy with the last dose within 14 days prior to Screening, or had a viral upper respiratory infection within 7 days prior to Screening;
* had asthma, unless their symptoms could be controlled by a short-acting inhaled Beta2-agonist used on an "as needed" basis;
* were on immunotherapy, unless they were on a stable maintenance schedule prior to screening. The dose of immunotherapy should remain constant and subjects could not receive immunotherapy within 24 hours prior to any visit;
* had a history of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that were likely to limit the validity of consent to participate in the study;
* had a history of non-compliance with medications or treatment protocols;
* had any clinically significant deviation from normal in the physical examination that, in the Investigator's judgment, may have interfered with the study evaluations or affect subject safety;
* had any clinically significant metabolic, cardiovascular, immunologic, neurologic, hematologic, gastrointestinal, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the Investigator, might interfere with the study evaluations or affect subject safety;
* had liver or renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2002-11-01 (Actual); Primary Completion 2003-06-01 (Actual); Study Completion 2003-06-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measure was the preference rates calculated from subject comparative evaluation. | 1 day after the end of each 7-day treatment period (Visit 3 and Visit 5)

SECONDARY OUTCOMES:
Subject Non-Comparative Evaluation and subject Response to Therapy | 1 day after the end of each 7-day treatment period (Visit 3 and Visit 5)